CLINICAL TRIAL: NCT01433471
Title: Mucosal Immunity of Ulcerative Colitis Patients Undergoing Therapy With Trichuris Suis Ova
Acronym: MUCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R#11-02470
Record Dates: First submitted 2011-09-06; First posted 2011-09-14 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Trichuris Suis Ova; Inflammatory Bowel Disease; Mucus
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trichuris suis ova followed by placebo (Experimental): Subjects in this arm will receive Trichuris suis ova for 12 weeks, followed by placebo for 12 weeks after crossover
  Interventions: Drug: Trichuris suis ova
- Placebo followed by Trichuris Suis Ova (Active Comparator): Subjects in this arm will receive placebo for 12 weeks, followed by Trichuris suis ova for 12 weeks after crossover
  Interventions: Drug: Trichuris suis ova

INTERVENTIONS:
Drug: Trichuris suis ova — 2,500 eggs by mouth every two weeks for 12 weeks
  Other Names: TSO

SUMMARY:
The purpose of this study is to understand the immune response activated in the human gastrointestinal tract by Trichuris Suis Ova (TSO) in patients with ulcerative colitis.

DETAILED DESCRIPTION:
The concept of helminthic therapy (using worms to treat diseases) is supported by experiments in mouse models as well as several clinical studies. TSO, which are purified eggs from the porcine whipworm Trichuris suis, are being investigated in clinical trials as a potential therapeutic agent for the treatment of active Crohn's disease, relapsing multiple sclerosis, peanut and tree nut allergy, and adults with autistic disorders.

The goal of this study is to understand the immune mechanisms activated in the human gastrointestinal tract by treatment with TSO, which may lead to improvements in the symptoms of ulcerative colitis (UC). TSO have been shown to have a clinical benefit on a subset of patients with UC in a previous randomized placebo-controlled trial (Summers et al. 2005). However, the mechanisms of action of TSO on the intestinal mucosa remain unclear.

We propose an exploratory 24-week mechanistic randomized double-blind placebo-controlled crossover study of TSO in patients with established and active UC to better characterize similarities and differences in the immune mechanisms of the intestinal mucosa in response to TSO. We hypothesize that treatment with TSO will lead to an anti-inflammatory immune response in some individuals with UC through an increase in intestinal mucus production and modulation of Th1, Th2, Th17, and T-regulatory effector lymphocyte populations.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be outpatients between the ages of 18 and 72.
* Subjects must have a biopsy-proven diagnosis of ulcerative colitis for greater than three months.
* There should be evidence of active disease with a total Mayo score of 6 to 10 points (scores range from 0 to 12, with higher scores indicating more severe disease activity).
* There should be moderate (marked erythema, lack of vascular pattern, friability, erosions) to severe (spontaneous bleeding, ulceration) active disease on colonoscopy (Mayo endoscopic score of at least 2) at time of enrollment.
* Laboratory inclusion criteria will require a hemoglobin level of >9.0 g/dL, a white blood count between 5,000 and 15,000/μL, a platelet count of >100,000μL, a blood urea nitrogen < 40mg/dL, a serum creatinine of <2.0mg/dL, a total bilirubin < 2.5 mg/dL, and an alkaline phosphatase of <250U/dL.
* Women will be required to have a negative urine pregnancy test and to practice birth control.
* The following medications will be allowed and continued throughout the study: Oral or rectal sulfasalazine, mesalamine, or mesalamine derivative (maintenance therapy of > 8 weeks, stable dose of > 4 weeks); Oral corticosteroid (prednisone, prednisolone, or budesonide) at an equivalent dose of a maximum of 40mg daily prednisone (maintenance therapy of >4 weeks, stable dose of > 2 weeks), azathioprine or 6-mercaptopurine (maintenance therapy of > 8 weeks, stable dose of > 4 weeks).
* Subjects must have the ability to provide informed consent and be willing to keep all scheduled appointments for the duration for the study period.

Exclusion Criteria:

* Inpatients, pregnant patients, patients with impaired cognition, patients with a history of active substance abuse in the past six months, and children.
* Patients with a history of bowel surgery in the prior six months or who currently or previously had an ileostomy or colostomy.
* Patients with active malignancy or treatment with anticancer drugs in the past 5 years, have a history of colorectal cancer or dysplasia, or a history of neoplasm of the gastrointestinal tract.
* Female patients who are pregnant, breastfeeding, wishing to become pregnant during study participation, or unwilling to use birth control.
* Patients with white blood count <5,000 or >15,000/mm3; platelet count <150,000 per μl; or iron or vitamin B12 deficiency. Correction of lab exclusion is allowed provided that medical condition is not deemed to put patient at risk and stability of result is sustained for a minimum of 30 days.
* Patients with stools positive for enteric pathogens, ova, or parasites at Screening
* Patients with active hepatitis B virus or hepatitis C virus infection or have been exposed to human immunodeficiency virus (HIV).
* Patients who have received an anti-tumor necrosis factor inhibitor (e.g. infliximab) within 12 weeks prior to Screening
* Patients who have received antibiotic, antifungal or antiparasitic medication in the last 2 weeks prior to Screening and/or would potentially require this during the study treatment period.
* Patients with evidence of poor compliance with medical advice and instruction including diet or medication.
* Patients who are unable or unwilling to swallow study medication suspension.
* Patients will be excluded if they have previously attempted helminthic therapy.
* There must not be evidence of fulminant colitis or a Mayo score of greater than 10
* Patients will be excluded if other clinically significant disease is present that could interfere with protocol compliance or interpretation of the results.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Poles, M.D., Ph.D., Principal Investigator — NYU Langone Health; P'ng Loke, Ph.D., Principal Investigator — NYU Langone Health; Martin J Wolff, M.D., Study Director — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trichuris Suis Ova Followed by Placebo | Placebo Followed by Trichuris Suis Ova
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trichuris Suis Ova Followed by Placebo | Placebo Followed by Trichuris Suis Ova | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of Mucus Production at 12 Weeks and 24 Weeks as Assessed by Histopathology
Time Frame: Baseline, 12 weeks, 24 weeks
Population: Because of the small sample size of this study, investigators decided it was not possible to draw meaningful conclusions from the outcome measures and outcome measures were not collected or analyzed as originally planned. Therefore, no outcome measure data is available.
Arm/Group | Trichuris Suis Ova | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change From Baseline of Effector Lymphocyte Populations (Th1, Th2, Th17, and T-regulatory Cells) at 12 and 24 Weeks as Assessed by Flow Cytometry of Peripheral Blood Mononuclear Cells and Isolated Leukocytes From Pinch Biopsies
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 1
Arm/Group | Trichuris Suis Ova Followed by Placebo | Placebo Followed by Trichuris Suis Ova
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change From Baseline of Bacterial Composition and Attachment at 12 Weeks and 24 Weeks as Assessed by Real-time Polymerase Chain Reaction and 454 Sequencing of Pinch Biopsies and Stool Specimens
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 1
Arm/Group | Trichuris Suis Ova Followed by Placebo | Placebo Followed by Trichuris Suis Ova
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Change From Baseline of Gene Expression at 12 Weeks and 24 Weeks as Assessed by Microarray and Real-time Polymerase Chain Reaction Analysis of Pinch Biopsies
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 1
Arm/Group | Trichuris Suis Ova Followed by Placebo | Placebo Followed by Trichuris Suis Ova
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Mayo Score From Baseline at 12 Weeks and 24 Weeks
Description: To assess ulcerative colitis disease activity
Time Frame: Baseline, 12 weeks, 24 weeks
Population: as for outcome 1
Arm/Group | Trichuris Suis Ova Followed by Placebo | Placebo Followed by Trichuris Suis Ova
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline of the Simple Clinical Colitis Activity Index at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24 Weeks
Description: To assess ulcerative colitis disease activity without requiring endoscopy
Time Frame: Baseline, 2, 4, 6, 8, 10, 14, 16, 18, 20, 22 weeks
Population: as for outcome 1
Arm/Group | Trichuris Suis Ova Followed by Placebo | Placebo Followed by Trichuris Suis Ova
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Trichuris Suis Ova | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trichuris Suis Ova (N=3) | Placebo (N=4)
Abdominal pain (General disorders) | 3 (4) | 3 (3)
Abdominal fullness (General disorders) | 2 (2) | 2 (2)
Excess flatulence (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Perianal pruritis (Gastrointestinal disorders) | 1 (2) | 2 (5)
Fatigue (General disorders) | 2 (2) | 2 (2)
Nausea/Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Increase in ALT (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Because of the small sample size of this study, investigators decided it was not possible to draw meaningful conclusions from the outcome measures and outcome measures were not collected or analyzed as originally planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No